CLINICAL TRIAL: NCT05187312
Title: Research Registry for Endoscopic Treatment and Diagnostics
Brief Title: Registry for Advanced Endoscopy
Acronym: ERDB
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-7616
Record Dates: First submitted 2021-12-25; First posted 2022-01-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Cholangiocarcinoma; Pancreatic Cancer; Sclerosing Cholangitis
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Cholangitis, Sclerosing | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, bile, tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic retrograde Cholangio- pancreatography — Endoscopic intervention in the biliary or pancreatic duct
Procedure: Endoscopic ultrasound — Endoscopic investigation/intervention with ultrasound

SUMMARY:
Observational registry including endoscopic diagnostic and therapeutic interventions in the gastrointestinal tract

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for endoscopic intervention/procedure

Exclusion Criteria:

* No informed consent
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for endoscopic procedures at Karolinska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2032-01-14 (Estimated); Study Completion 2032-01-14 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 30-days and 60-days post-procedure
  Incidence of Adverse events following endoscopic procedures. Measured as percentage of individuals with an adverse event
Diagnostic yield | 1-year follow up
  Diagnostic yield after tissue sampling

CONTACTS AND LOCATIONS:
Overall Officials: Erik von Seth, MD, PhD, Principal Investigator — Region Stockholm
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No